CLINICAL TRIAL: NCT02126930
Title: Impact of a Pharmaceutical Consultation at Hospital Discharge on Adherence to Anti-infective Treatment After Returning Home
Brief Title: Pharmaceutical Consultation at Hospital Discharge and Adherence to Anti-infective Treatment
Acronym: CPS-INFECTIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2014/HF-01; 2014-A00335-42 (Other: RCB number); 2014-A00944-43 (Other: RCB number); LOCAL/2014/AS-01 (Other: obsolete sponsor number)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Infection
Keywords: anti-infectious treatment; observance; pharmaceutical consultation
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine care (Active Comparator): The patients in this receive routine care.
  Intervention: Routine care
  Interventions: Other: Routine care
- Pharma consult (Experimental): The patients in this arm will have a pharmaceutical consult upon hospital discharge.
  Intervention: Pharma consult
  Interventions: Other: Pharma consult

INTERVENTIONS:
Other: Pharma consult — Upon hospital discharge, patients randomized to the experimental arm will have a pharmaceutical consultation concerning their anti-infectious treatment.
  Arms: Pharma consult
Other: Routine care — Patients randomized to this arm will receive care in the habitual manner.
  Arms: Routine care

SUMMARY:
The main objective of this study is to evaluate the impact of a pharmaceutical consultation at the time of hospital discharge on the adherence of patients ; non-adherence is determined by the following criteria:

As concerns prescribed anti-infectious treatments, at least one of the following 4 criteria is true:

1. . the patient did not go and get his/her treatment at the pharmacy;
2. . the number of treatment units dispensed by the pharmacy is < the number of treatment units prescribed;
3. . the patient stopped taking a treatment before the recommended time, or continued taking a treatment after the recommended time;
4. . the number of treatment units taken by the patient (self-declaration) is < or > to the number of units prescribed.

DETAILED DESCRIPTION:
The secondary objectives of this study are :

A- To assess the percentage of patients who obtained their anti- infective pharmaceuticals

B- To evaluate the ratio of the number of units of anti- infective drugs dispensed by the pharmacy over the number of units of anti- infective drugs prescribed

C- To determine the ratio of the number of premature discontinuations of anti -infective treatments over the number of lines of anti -infective treatments prescribed

D- Evaluate the ratio of the number of units actually taken by the patient (based on a self-declaration) over the number of units of anti- infective drugs prescribed

E- To measure the comprehension concerning anti- infective treatments after returning home (based on a quiz)

F- To determine the risk factors for non- adherence to anti- infective therapy based on the characteristics of the study population

G- Assess patient satisfaction concerning a pharmaceutical consultation at hospital discharge (questionnaire)

H- Assess the impact of a pharmaceutical consultation on primary non-adherence (criteria 1 and 2) and secondary non- adherence (criteria 3 and 4)

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is hospitalized in the Infectious and Tropical Diseases department of the Nîmes University Hospital, and is scheduled for hospital discharge with one or more pharmaceutical prescriptions for anti-infectious treatments

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient resides in a care establishment, or has home medical/nursing service
* The patient is suffering from chronic infection (>4 weeks of treatment required)
* The patient is suffering from handicapping deafness, dementia, or does not have a telephone
* Intravenous, intramuscular or subcutaneous anti-infectious treatments are prescribed
* Prescription of antiretroviral treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The presence/absence of treatment non-adherence | 1 week after end of treatment (expected max of 4 weeks)
  As concerns prescribed anti-infectious treatments, at least one of the following 4 criteria is true:
  1. . the patient did not go and get his/her treatment at the pharmacy;
  2. . the number of treatment units dispensed by the pharmacy is < the number of treatment units prescribed;
  3. . the patient stopped taking a treatment before the recommended time, or continued taking a treatment after the recommended time;
  4. . the number of treatment units taken by the patient (self-declaration) is < or > to the number of units prescribed.

SECONDARY OUTCOMES:
Delivery of anti-infectious therapy by the pharmacy (yes/no) | 1 week after end of treatment (expected max of 4 weeks)
Number of anti-infectious drug units dispensed by the pharmacy / number of anti-infections drug units prescribed | 1 week after end of treatment (expected max of 4 weeks)
Number of premature discontinuations of anti-infective therapies / the prescribed number of anti-infective treatments | 1 week after end of treatment (expected max of 4 weeks)
Number of anti-infectious drug units taken by the patient (self-declaration) / number of anti-infections drug units prescribed | 1 week after end of treatment (expected max of 4 weeks)
Quiz on anti-infective therapy comprehension | Day 0 (hospital discharge)
Socio-demographic characteristics | Day 0 (hospital discharge)
Test for measuring overall compliance (MAQ) | Day 0 (hospital discharge)
Satisfaction Questionnaire concerning pharmaceutical consultation | Day 0 (hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Harmonie Faure, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France